CLINICAL TRIAL: NCT00088348
Title: Screening Study for the Evaluation and Diagnosis of Potential Research Subjects With Anterior Segment Disease
Brief Title: Screening for Research Subjects With Anterior Segment Diseases
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040241; 04-EI-0241
Record Dates: First submitted 2004-07-23; First posted 2004-07-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-08-20

CONDITIONS: Eye Diseases
Keywords: Cornea; Conjunctiva; Keratitis; Ocular Surface; Inflammation; Evaluation; Screening; Ocular Surface Disease; Eye; Ocular Disease; Anterior Segment Disease
MeSH Terms: conditions — Eye Diseases; Corneal Diseases; Keratitis; Inflammation

SUMMARY:
This study will identify patients with anterior segment disease who may be eligible to participate in current or future NEI studies on this disease. Anterior segment disease includes all disorders that affect the eye surface, anterior chamber, iris and ciliary body and lens of the eye. The eye surface is composed of the cornea, conjunctiva, eyelids, lacrimal and meibomian glands, and the interconnecting nerves.

Patients of any age with anterior segment disease may be eligible for this screening study. Participants will be evaluated with some or all of the following tests and procedures, depending on the nature of their eye problem:

* Medical history and brief physical examination.
* Eye examination, including measurement of visual acuity (eye chart) and eye pressure, examination of the pupils, eye movements, structures in the front of the eye (cornea, conjunctive, etc.), the lens, and the structures in the back of the eye (retinal, optic nerve, etc.).
* Photographs of the eye to help assess the status of the cornea and conjunctive and to evaluate any changes that may occur in the future.
* Assessment of tear and surface status. The amount of tears the eyes can produce is measured by placing a small piece of sterile paper in the corner of the eye every 5 minutes. Special orange and green dyes are placed in the eyes to determine the health status of the surface of the eye.
* Corneal or conjunctival biopsy. A small tissue sample from the surface of the eye may be removed for laboratory examination to help diagnose a condition that is unclear. For this procedure, the eye is numbed with anesthetic eye drops. The required tissue is collected, an antibiotic ointment is placed in the eye to prevent infection, and a patch may be placed over the eye for 12 to 24 hours.
* Blood draw for tests to study the cause of the patient's eye disease.
* Other diagnostic tests as needed.
* DNA testing to look for a genetic pattern associated with the patient's eye disease.

Patients who are found eligible for an NEI study will be offered participation in that study. Patients who are not eligible for current studies will be advised about treatment options.

DETAILED DESCRIPTION:
This is a screening protocol that will allow the NEI clinicians to examine patients with ocular diseases in order to identify those who may be eligible to participate in other NEI studies on anterior segment disease.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

To participate in this screening study, a patient must have a history of anterior segment disease. Patients of all ages are eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 2004-07-13; Study Completion 2008-08-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Holland EJ. Epithelial transplantation for the management of severe ocular surface disease. Trans Am Ophthalmol Soc. 1996;94:677-743. PMID 8981714